CLINICAL TRIAL: NCT04345653
Title: Feasibility, Safety and Early Efficacy Trial of Hydroxychloroquine as Primary Prevention of Corona Virus Disease 2019 in High Risk Health Care Providers
Brief Title: Hydroxychloroquine as Chemoprevention for COVID-19 for High Risk Healthcare Workers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2020-0356
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: covid19; workers; prevention
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm - Hydroxychloroquine Sulfate (HCQ) (Experimental): HCQ sulfate HCQ 400mg (2x 200mg tablets) by mouth 6-12 hours apart on day 1, followed by 3 weeks of weekly 400mg (2x 200mg tablets) by mouth
  Interventions: Drug: Hydroxychloroquine Sulfate (HCQ)

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate (HCQ) — Open-label, consecutive at-risk subjects allocation with chemoprophylaxis with HCQ.

SUMMARY:
The study proposes to conduct an open-label Phase II trial to evaluate the feasibility, safety and early efficacy of hydroxychloroquine (HCQ) administration in reduction of transmission of severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) and development of Corona Virus Disease 2019 (COVID-19) in high-risk, healthy acute care provider participants exposed, directly or indirectly, to COVID-19 patients. There is a more than 50 years track record of safety of HCQ for treatment and prevention of various disease states. Early data on use of HCQ for COVID treatment suggests anti-viral activity and immunomodulatory properties for reducing inflammation associated with COVID-19.

DETAILED DESCRIPTION:
Given the lack of data regarding use of HCQ for COVID-19 prevention in healthy participants in midst of pandemic crisis, this study proposes an expedited feasibility study focusing on safety and early efficacy.

Prior to HCQ administration, baseline SARS-CoV-2 and other baseline biomarker testing will be conducted. During the 4-week study period, participants will be monitored for drug related adverse events and assessed for development of COVID. SARS-CoV-2 assay and biomarker testing will be repeated at the end of four-week study. Safety outcomes will be assessed by the number of adverse events (AEs) and their severity; and early efficacy as the number of participants who tested positive at the end of the 4-week period comparing to data collected by occupational Health regarding the total number of high-risk healthcare workers that were tested positive during the same period and historical controls from known high risk infection rates. An exploratory analysis of inflammatory regulation and immunomodulatory markers by HCQ and its effect on possible disease modification based on previously studied pathophysiological mechanism of COVID-19.

The broader aim of this study is to set a precedent to facilitate a large-scale emergent public health intervention. Purpose would be to mitigate, or abort further transmission of COVID-19. Given that COVID-19 transmission has occurred prior to initiation of this study, the rationale for this intervention is based on prior epidemiological evidence. Post-infectious or vaccination-induced immunity in at least 30% of population at-risk has been shown to mitigate or abort propagation of a local epidemics and global pandemic. This would help flatten the curve of the disease progression, until such time that a vaccine may become available. Data from this study will be used to design and implement a population-based phase IIb/III randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers ages 18 to 99 years,
* Able to sign own informed consent form,
* Considered high-risk healthcare care providers in a hospital setting with active exposure to COVID-19 infection.

High-risk healthcare providers are defined as those actively working during the study duration in the Emergency Department and in the Intensive Care Setting, for the purpose of this study.

Exclusion Criteria:

* Inability to tolerate an oral medication or known allergy to chloroquine or hydroxychloroquine
* Pregnancy or breast-feeding
* Immunocompromised status, hepatic failure, electrolytic imbalance
* Creatinine clearance (CCL) <30 mL/min
* Prolonged QT interval (QTc > 450ms for males and QTc > 470 for females)
* Confirmed COVID-19 infection on baseline testing
* Has another known contraindication to treatment with the study drug, including retinopathy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jawad Kirmani, MD, Principal Investigator — Hackensack Meridian Health Corporation
Locations (1):
- Hackensack Meridian Health - JFK Medical Center, Edison, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Arm - Hydroxychloroquine Sulfate (HCQ)
Started | 48
Completed | 46
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: High risk healthcare providers
Arm/Group | Study Arm - Hydroxychloroquine Sulfate (HCQ)
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 39.5 [26.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility
Description: To evaluate the feasibility of this protocol including participants' recruitment within the estimated time frame, i.e. understand the ability of the team to identify eligible participants, enroll them, retain them and follow them up until study completion.
Time Frame: Study period, up to two months from the day the first participant was screened
Population: High risk healthcare providers
Measure: Count of Participants; unit: Participants
Groups:
- Study Arm: HCQ sulfate HCQ 400mg (2x 200mg tablets) by mouth 6-12 hours apart on day 1, followed by 3 weeks of weekly 400mg (2x 200mg tablets) by mouth
  Hydroxychloroquine Sulfate (HCQ): Open-label, consecutive at-risk subjects allocation with chemoprophylaxis with HCQ.
Arm/Group | Study Arm
Number analyzed (Participants) | 46
Participants | 46

2. Primary Outcome: Resource Utilization
Description: To evaluate the utilization of tests and drug for this study in consideration with the limited availability of both for research purposes as reflected on the number of participants that got tested and received at least one dose of the drug.
Time Frame: Study period, up to two months from the day the first participant was screened
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Hydroxychloroquine Sulfate (HCQ)
Number analyzed (Participants) | 46
Participants | 46

3. Primary Outcome: Safety as Reflected on the Number and Severity of Adverse Events and Serious Adverse Events
Description: To Determine the Safety profile for a previously well studied drug in this select group of HCP. Incidence of well described side effects would be studied over the course of the study and will be compared with the side effects and their prevalence as described in the Pharmacy manual for HCQ.
Time Frame: 28 day post enrollment
Population: High risk healthcare providers
Measure: Number; unit: Adverse Events
Arm/Group | Study Arm - Hydroxychloroquine Sulfate (HCQ)
Number analyzed (Participants) | 46
Adverse Events
  Serious Adverse events | 0
  Adverse events | 24

4. Primary Outcome: Early Feasibility as Reflected on the Number of Participants Contracting COVID-19 (10% or Less) in Comparison to the Expected 30% as Per CDC.
Description: To evaluate the early efficacy of HCQ in high-risk, healthy volunteers in the prevention of acquiring COVID-19 while continuing to follow standard precautions that meet or exceed Centers of Disease Control (CDC) guidelines.
Time Frame: 28 day post enrollment
Measure: Number; unit: participants
Arm/Group | Study Arm - Hydroxychloroquine Sulfate (HCQ)
Number analyzed (Participants) | 46
participants | 0

ADVERSE EVENTS:
Time Frame: Overall follow up period: 6 month
Arm/Group | Study Arm - Hydroxychloroquine Sulfate (HCQ)
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 24/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm - Hydroxychloroquine Sulfate (HCQ) (N=46)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Headaches (Nervous system disorders) | 3 (3)
Shortness of breath and chest pain (Cardiac disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Mood Disorder (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT04345653/Prot_SAP_000.pdf